CLINICAL TRIAL: NCT05062512
Title: Health in Aging, Neurodegenerative Diseases and Dementias In Ontario
Acronym: HANDDS-ONT
Status: Terminated | Type: Observational
Why Stopped: Funding not renewed.
Sponsor: Ontario Neurodegeneration Disease Research Initiative (Other)
Collaborators: Ontario Brain Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 3589
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Neuro-Degenerative Disease; Dementia
Keywords: observational; remote; wearable technology; genomics
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collected samples (serum, plasma, DNA, RNA) will be used for analyses including, but not limited to:
  * total tau protein, phosphorylated tau-181 (p-tau181), neurofilament light chain (NfL), glial fibrillary acidic protein (GFAp), Neuron-specific enolase (NSE), S100 calcium-binding protein B (S100B), amyloid beta 40 and 42 (AB-40, AB-42), alpha-synuclein markers.
  * additional emerging approaches (e.g. lipidomics, RNA analysis) help to understand processes of aging, vascular risk, inflammation and other factors that can accelerate decline and/or promote health.
  * whole genome sequencing will be performed to identify potential genetic variants that may predict underlying neurodegenerative disease and dementia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants living with and without neurodegenerative diseases: No intervention

SUMMARY:
The Health in Aging, Neurodegenerative Diseases and DementiaS in ONTario (HANDDS-ONT) Study is an observational study that takes place in the comfort of participant's home, with no study visits occurring in a clinic. The study is recruiting people living with a neurodegenerative disease or the effects of stroke, along with healthy, aging individuals. Studying both groups will help ONDRI researchers to:

1. understand how the diseases affect different people
2. discover ways to potentially detect diseases earlier
3. find ways to help people manage their daily health related behaviours

Participant data is collected virtually through wearables - small sensors worn on the wrist, ankle and chest -- for 7-10 days, as participants go about their daily activities. Data is also collected from questionnaires regarding mood and quality of life. Blood samples will be collected to understand how one's genetic makeup could provide for earlier detection of some conditions, and for analysis of certain risk factors. Combining the information from the sensors (walking patterns, sleep, heart rate/rhythm, etc.), the questionnaires and the blood samples will allow researchers to better understand aging, with and without a neurodegenerative condition, over a period of time.

Participants will receive a personalized health and activity report, describing sleep and activity during the time the wearable sensors were worn. This information may help participants better understand and manage some aspects of their overall health and it can be shared with their circle of care.

DETAILED DESCRIPTION:
HANDDS-ONT is designed with the following principal research question in mind:

Can the integration of biosamples, clinical data and remote wearable biosensor data across aging and neurodegenerative disease cohorts i) provide valuable diagnostic data, ii) demonstrate predictive utility for important clinical outcomes and iii) guide daily decisions and care for individuals living with neurodegenerative diseases? Ultimately we aim to improve the lived-experience of individuals affected by dementia. This protocol focuses on building the foundation for this long-term objective by adapting the NIA-AA framework to link genetic, proteomic, and free-living behavioural signatures across NDD cohorts.

Objectives:

Objective 1 will examine the expression of single proteins or sets of proteins (i.e., protein biomarkers), and different gene mutation inheritance patterns (e.g. mutation negative, monogenic mutation, polygenic mutations), to help identify unique cohorts with similar symptoms and free-living behavioural profiles.

Objective 2 will examine the relationship between multidimensional data (genomic-proteomic signatures, functional behaviours extracted from free-living data collected with wearable biosensors), and the risk for adverse health outcomes (e.g., ED visits, hospitalizations, long-term care admission, death, comorbid disease).

Objective 3 will examine the useability, acceptance and impact of feedback on self-management activities. Feedback around functional activities will be provided in the form of a participant report that conveys higher level metrics intended to inform and/or alter behavior relative to overall health, symptom management, and/or quality of life.

HANDDS-ONT is designed as a "Master Observational Trial" [https://doi.org/10.1016/j.cell.2019.12.009], connecting real-world clinical data with cellular, protein marker and genetic data, free-living behavioural data measured by wearable biosensors and longer-term health outcome data via linkage to administrative datasets at ICES.

Data collection will build on existing ONDRI research infrastructure and a central group of research cores that reflect the evolving state of research in neurodegenerative disorders. Specifically, there will be five complimentary research cores (Fluid biomarkers, Clinical, Wearable biosensors, Health Systems, and Neuroinformatics) overseen by a central research Administration Core.

To achieve Objective 1, fluid biomarkers from serum and plasma, genetic data, clinical information and free-living behaviours (e.g. sleep, physical activity and other markers collected using wearable biosensors) will be integrated to identify groups based on NIA-AA research framework. Participants will be asked to provide a blood sample, complete standardized questionnaires for data collection by telephone or online, and wear wearable biosensors for 7-10 days described in sections below.

To achieve Objective 2, the clinico-pathological cohorts identified in objective 1 (combining protein and genetic biomarker data with clinical and free-living behaviour data) will be linked to administrative datasets at ICES to identify risk factors for important clinical outcomes (e.g. death, long-term care need, comorbid diseases, falls) and patterns of health systems utilization. Participants will be asked for permission to securely store Health Card Numbers and link to ICES for outcomes (see Procedures and Assessments section, below).

To achieve Objective 3, surveys and interviews will be administered. As additional metrics are validated, they will be integrated into the feedback form for evaluation using the methods described in Objective 3, above. Participants may consent to being recontacted for ongoing feedback and new study options (see Procedures and Assessments section, below).

ELIGIBILITY:
Inclusion Criteria:

* All Participants:

  1. Informed Consent provided by participant or substitute decision maker
  2. Age 18 and older
  3. Participant must rate his/her level of proficiency speaking and understanding English at 7 out of 10 or higher on the a modified version of the LEAP-Q *
  4. Telephone or internet access
  5. Ability to attend a LifeLab facility of participant's choice to provide blood sample
  6. Under the care of a primary medical care provider (e.g. family physician or nurse practitioner) and/or specialist and their name provided for purposes of reporting incidental findings.

     * Participants must have proficiency in English to understand study instructions and respond to questionnaires licensed for use in English only. Study does not have resources for translation of study documents/certified translators.

Participants with Neurodegenerative Diseases:

1. Participant-reported diagnosis of meeting "possible or probable" clinical criteria for AD, MCI, PD, PD+ (e.g. MSA/PSP/CBD/LBD), ALS, FTD or Cerebrovascular disease.
2. Aging adults without a specific diagnosis, but who have cognitive symptoms (Telephone Interview for Cognitive Status-Modified (TICS-M; Total score <32) will be assigned to the MCI cohort.

Exclusion Criteria:

* Underlying conditions which may interfere with the participant's ability to participate in the study or may compromise study results, including but not limited to:

  1. Contraindication to the biosensors as outlined by biosensor manufacturers,
  2. Substance abuse within the past year or history of alcohol or drug abuse which the study team feels may interfere with the participant's ability to comply with the study procedures.
  3. Known brain tumour (e.g. glioblastoma, metastatic cancer to the brain)
  4. Prior brain surgeries that the study team feels will interfere with participation
  5. Known history of poor venous access or difficulties with blood draws
  6. Significant psychiatric disorders (e.g. untreated major depression, psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 500 participants from multiple groups will be recruited: those with diagnoses of neurological disorders associated with neurodegeneration and increased risk for dementia (e.g., PD, MCI/AD, cerebrovascular injury +/- cognitive impairment, ALS, Fronto-temporal dementia) as well as healthy adult aging controls
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Generate behavioural/functional profiles from the wearable biosensors | 7-10 day sensor wear period
  data collected during the biosensor wear period will be post-processed to extract additional summary measures and patterns of behaviour. Sample measures include: amount of time in sedentary/light/moderate/vigorous intensity activity, total active minutes, estimate of energy expenditure, total walking activity, step count, walking bout durations, characteristics of walking (e.g. cadence, gait velocity, etc.), imbalance and fall events, sleep duration, number of arousals, inter-daily sleep stability, intra-daily sleep variability, sleep fragmentation, heart rate (beats per minute), heart rate variability.
identify profiles of clinical and functional expression | 2 years
  a semi-guided approach will identify multivariate projections using techniques such as PCA and CA from summary measures with prima facie validity of association with cognition (e.g. variability of cardiac RR interval, average total sleep time, first quartile of Fourier transform of acceleration while walking, body mass index, age) extracted from clinical eCRF and biosensor data streams.
select subsets of genomic and proteomic features | 2 years
  . Multiple (mass) univariate tests will be used to rank features and false discovery rate adjustment will be used to establish feature selection threshold. Identification of multivariate associations will be performed by simultaneous models of the independent projections on the multiple genomic-proteomic features with penalized optimization. Multi-class LASSO or sparse LDA will be used to identify features associated with clinical-functional clusters.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Swartz, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected for the purpose of publications are to be shared via a controlled public release along with accompanying data dictionaries and other supplementary files. All data share are de-identified in accordance with the policies set out by the Ontario Brain Institute (OBI).
Time Frame: Data will be released in the future and available with supporting information per OBI's guidelines.
Access Criteria: Access to data is provided to users with an affiliation with an accredited academic institution, think tank, company, or other research organization. Users must also submit a Data Access Request along with Research Ethics Board approval which are then reviewed and approved by OBI's data access committee.
URL: https://indocconsortium.atlassian.net/wiki/spaces/JSDNXT/pages/1933279255/Data+Release+Articles